CLINICAL TRIAL: NCT01469923
Title: A Phase I, Single Centre, Single-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD2820 After Administration of Multiple Ascending Doses
Brief Title: To Assess the Safety, Tolerability, Pharmacokinetics and Pharmakodynamics of AZD2820 After Multiple Ascending Doses
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D3870C00002
Record Dates: First submitted 2011-09-30; First posted 2011-11-10 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Obesity
Keywords: Phase 1; obese; healthy male volunteers; multiple doses; dose escalation; pharmacokinetics; pharmakodynamics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- AZD2820 (Active Comparator): AZD2820 multiple injections
  Interventions: Drug: AZD2820
- Placebo for AZD2820 (Placebo Comparator): Placebo for AZD2820 multiple injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2820 — Ascending subcutaneous injections of AZD2820 once daily for 14 days in the abdomen
  Arms: AZD2820
Drug: Placebo — Ascending subcutaneous injections of placebo for AZD2820 once daily for 14 days in the abdomen
  Arms: Placebo for AZD2820

SUMMARY:
This is a randomised and single-blind, placebo-controlled study to investigate the safety, tolerabilty, pharmacokinetics and pharmacodynamics of repeated and ascending doses of AZD2820 to obese but otherwise healthy male subjects.

DETAILED DESCRIPTION:
A Phase I, Single Centre, Single-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD2820 after Administration of Multiple Ascending Doses.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures including the genetic sampling and analyses
* Obese but otherwise healthy male subjects aged 18 - 45 years with suitable veins for cannulation or repeated venepuncture
* Male subjects should be willing to use barrier contraception ie, condoms, from the first day of dosing until 3 months after the last dose of investigational product
* Have a body mass index (BMI) between 27 and 40 kg/m2

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the stud
* A history of erectile dysfunction or anatomic abnormality of the penis (eg, cavernosal fibrosis, Peyronie's disease, or plaques) which interferes with normal erectile function
* Prolonged QTcF >450 ms or shortened QTcF <340 ms or family history of long QT syndrome
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD2820
* Any clinically significant abnormalities in clinical chemistry, haematology (including eosinophilia) or urinalysis results as judged by the investigator

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Description of the safety and tolerability profile of AZD2820 in terms of adverse events. | From baseline, defined as day 1 of dosing, up to day 29
  No formal statistical test will be performed. Abnormalities will be listed without statistical analysis.
Description of the safety and tolerability profile of AZD2820 in terms of labolatory data ( clinical chemistry, haematology and urinalisys). | From baseline, defined as one day prior first dose, up to day 28.
  No formal statistical test will be performed. Abnormalities will be listed without statistical analysis.
Description of the safety and tolerability profile of AZD2820 in terms of vital signs ( pulse, systolic and diastolic blood preassure ( SBP, DBP and 24h ambulatory BP), body temperature). | From baseline, defined as one day prior first dose, up to day 29.
  No formal statistical test will be performed. Abnormalities will be listed without statistical analysis.
Description of the safety and tolerability profile of AZD2820 in terms of total immunoglobulin levels. | From baseline, defined as one day prior first dose, up to day 44.
  Number of subjects with immunoglobuline level outsite of reference range. No formal statistical tests will be performed. Abnormalities will be listed without statistical analysis.
Description of the safety and tolerability profile of AZD2820 in terms of safety electrocardiogram (ECG). | From baseline, defined as last pre dose measurement, up to day 28.
  No formal statistical test will be performed. Abnormalities will be listed without statistical analysis
Description of the safety and tolerability profile of AZD2820 in terms of digital electrocardiogram (ECG). | From baseline, defined as assessment at screening visit and day 1 of dosing.
  No formal statistical test will be performed. Abnormalities will be listed without statistical analysis. The QT correction factor will be based on the Fridericia's formula.
Description of the safety and tolerability profile of AZD2820 in terms of electroencephalography (EEG). | From baseline, defined as mean value of the 10 minutes recording prior first dose up to 7th day of dosing.
  No formal statistical test will be performed. Abnormalities will be listed without statistical analysis.
Description of the safety and tolerability profile of AZD2820 in terms of Columbia-Suicide Severity Rating Scale (C-SSRS). | From baseline, defined as one day prior first dose, up to day 12th of dosing.
  No formal statistical test will be performed. Abnormalities will be listed without statistical analysis.
Description of the safety and tolerability profile of AZD2820 in terms of skin pigmentation. | From baseline, defined as one day before first dose, up to day 29.
  No formal statistical test will be performed.
Description of the safety and tolerability profile of AZD2820 in terms of Penile erection (measured by Rigiscan). | From baseline, defined as one day before first dose, up 12th day of dosing.
  No formal statistical test will be performed.
Description of the safety and tolerability profile of AZD2820 in terms of physical examination. | From baseline, defined as two days prior first dose, up to day 29.
  No formal statistical test will be performed. Abnormalities will be listed without statistical analysis.

SECONDARY OUTCOMES:
Change in total caloric intake from baseline. | From baseline, defined as one day prior first dose to end of treatement which is day 15.
  Change from baseline will be measured after each meal and then grafically presented.
Description of the PK profile of AZD2820 in terms of Cmax, AUC(0-tau), AUC(0-t), AUC, (t1/2lz, h). | Day 1, PK samples collected post-dese at 20 min, 40 min, 1hr, 1.20hr, 1.40hr, 2hrs, 3hrs, 4hrs, 6hrs, 8hrs, 12hrs, 18hrs and 24hrs.
  Maximum drug plasma concentration (Cmax), Area under the drug plasma concentration-time curve from zero to the end of the dosing interval (AUC(0-tau), Area under the plasma concentration-time curve from zero to the time of the last quantifiable concentration (AUC(0-t)), Area under the plasma concentration time curve from zero to infinity (AUC), Terminal half-life (t1/2lz, h).
Description of PK profile of AZD2820 in terms of (Css,max, nmol/L), AUCss,(0-tau), (t1/2lz). | Day 7, PK samples collected post-dese at 20 min, 40 min, 1hr, 1.20hr, 1.40hr, 2hrs, 3hrs, 4hrs, 6hrs, 8hrs, 12hrs, 18hrs and 24hrs.
  Maximum plasma concentration at steady state (Css,max, nmol/L), Area under the plasma concentration-time curve from zero to the end of the dosing interval at steady state (AUCss,(0-tau)), Terminal half-life (t1/2lz).

CONTACTS AND LOCATIONS:
Overall Officials: James Ritter, BM BCH, MRCP, FRCP, Principal Investigator — QLON; Mark Berner Hansen, PHD, Study Director — AstraZeneca Mölndal, Sweden; Mirjana Kujacic, PHD, Study Chair — AstraZeneca Mölndal, Sweden
Locations (1):
- Research site, London, United Kingdom